CLINICAL TRIAL: NCT03973918
Title: A Phase II Study of Binimetinib in Combination With Encorafenib in Adults With Recurrent BRAF V600-Mutated High-Grade Astrocytoma or Other Primary Brain Tumor
Brief Title: Study of Binimetinib With Encorafenib in Adults With Recurrent BRAF V600-Mutated HGG
Acronym: BRAF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NCI decided to terminate ABTC Consortium due to NCI moving in different direction for Brain Cancer
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABTC 1802; UM1CA137443 (NIH)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: High Grade Glioma; BRAF V600E; BRAF V600K; Anaplastic Astrocytoma; Anaplastic Pleomorphic Xanthoastrocytoma; Gliosarcoma; Glioblastoma
Keywords: BRAF V600E/K; High Grade Primary Brain Tumor; High Grade Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Gliosarcoma; Glioblastoma | interventions — encorafenib; binimetinib; Circulating Tumor DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Cohort 1 AA & GBM (Experimental): Encorafenib 450mg QD Binimetinib 45mg BID 28 day cycle
  Research Bloods
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Biological: Research Bloods; Biological: Tumor Tissue
- Treatment Cohort 2 anaplastic PXAs (Experimental): Encorafenib 450mg QD Binimetinib 45mg BID 28 day cycle
  Research Bloods
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Biological: Research Bloods; Biological: Tumor Tissue
- Surgical Arm (Experimental): Pre-op -14 days: Encorafenib 450mg QD and Binimetinib 45mg BID last dose of both drugs 2hrs prior to surgery
  Tumor; research blood; CSF samples
  post surgery: Encorafenib 450mg QD Binimetinib 45mg BID 28 day cycle
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Biological: Research Bloods; Biological: Tumor Tissue
- Treatment Cohort 3 Other Tumors (Experimental): Encorafenib 450mg QD Binimetinib 45mg BID 28 day cycle
  Research Bloods
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Biological: Research Bloods; Biological: Tumor Tissue

INTERVENTIONS:
Drug: Encorafenib — 450mg QD 28 day cycle
  Other Names: Braftovi
Drug: Binimetinib — 45mg BID 28 day cycle
  Other Names: Mektovi
Biological: Research Bloods — Baseline; pre-cycle 3; Pre-cycle 7; off Treatment
  Other Names: Circulating Tumor DNA
Biological: Tumor Tissue — at time of surgery contrast enhancing and non enhancing tumor; 20 unstained slides

SUMMARY:
The goal of this study is to estimate the efficacy of encorafenib and binimetinib as measured by radiographic response in recurrent high-grade primary brain tumors.

DETAILED DESCRIPTION:
Primary Objective Estimate the efficacy of combination treatment with encorafenib and binimetinib, as measured by response rate (RANO criteria), in patients with recurrent BRAF V600E/K-mutated malignant glioma (MG) and anaplastic pleomorphic xanthoastrocytoma (PXAs).

Secondary Objectives

1. Estimate efficacy as measured by progression-free survival in subjects with recurrent malignant glioma or anaplastic PXA containing a BRAF-V600E/K mutation who receive drug.
2. Evaluate duration of response in subjects who have a partial or complete response.
3. Quantify the time-to-response among subjects who have a radiologic response.
4. Estimate efficacy as measured by overall survival in subjects with recurrent malignant glioma or anaplastic PXA containing a BRAF-V600E/K mutation who receive drug.
5. Characterize the toxicity profile of the combination of encorafenib and binimetinib in this patient population.

There are two arms: medical and surgical. Subjects on the surgical arm must have a high-grade glioma or a known BRAF-mutated low-grade glioma with high clinical suspicion for progression to high-grade.

Medical: Following enrollment, patients will receive encorafenib and binimetinib at the FDA-approved dose of 450 mg of encorafenib once daily and the FDA-approved dose of 45 mg of binimetinib twice daily separated by 12 hours, continuously in 28-day cycles until progression or unacceptable toxicity. Patients will be followed by routine blood work, and general and neurological examination. A brain MRI will be performed prior to every odd-numbered cycle (every 8 weeks). Response will be assessed by RANO criteria. Patients may remain on study and receive treatment until progression or other reason.

Surgical: These subjects will take encorafenib and binimetinib in combination at their FDA-approved doses for 10-14 days prior to surgery. The last dose of both drugs will be administered two hours prior to surgery. Specimens will be collected during surgery. After surgery, the subjects will not take further encorafenib or binimetinib until a study visit to assess their neurological exam, physical exam, and performance status, at 2-6 weeks post-operatively. At time of restarting combination treatment, subjects will follow the schedule for the medical cohort, and will continue treatment until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving any other standard or investigational agents are ineligible.
2. Patients with history or current evidence of the following conditions are excluded: neuromuscular disorder with associated elevated CK (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy), pancreatitis, retinal vein occlusion, uncontrolled HIV, or Hepatitis B/C. An exception will be made for (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months and for subjects with cleared HBV and HCV infections, who may enroll in the study.
3. Patients must have measurable (defined by at least 1 cm x 1 cm) contrast-enhancing disease by MRI imaging within 30 days of starting treatment.
4. The following intervals from previous treatments are required to be eligible:

   * 12 weeks from the completion of radiation.
   * 16 weeks from an anti-VEGF therapy
   * 4 weeks from a nitrosourea chemotherapy
   * 3 weeks from a non-nitrosourea chemotherapy
   * 2 weeks or 5 half-lives from any investigational (not FDA-approved) agents
   * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.)
5. Patients must be 18 years of age or older.
6. Patients must have a Karnofsky Performance (KPS) Status ≥ 60%
7. Patients must have adequate organ and marrow function within 30 days of starting treatment.
8. Patients must be able to provide written informed consent.
9. Women of childbearing potential must have a negative serum pregnancy test prior to study start. Women of childbearing potential must agree to use adequate contraception (intrauterine device, barrier, or other non-hormonal method of birth control; or abstinence) and not to donate ova from screening through 30 days after the last dose of study drug. Male participants must also agree to use adequate contraception and not to donate sperm from screening until 90 days after the last dose of study drug.
10. Patients must be maintained on a stable or decreasing dose of systemic corticosteroid regimen (no increase for 5 days) prior to baseline MRI. Topical and inhaled steroid treatment is allowed.
11. Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with other malignancies must be disease-free for ≥ 2 years.
12. Patients must be able to swallow tablets and capsules.
13. Patients must have a tumor tissue form completed and signed by a pathologist (see Section 9.6.4). The tumor tissue form must indicate availability of archived tissue. The archived tissue should be from the most recent tumor resection, demonstrating active tumor when sufficient tissue is available. If sufficient tissue is not available from the most recent surgery, then tissue from an earlier surgery is acceptable, if available, including from the initial resection at diagnosis.

Exclusion Criteria:

1. Patients receiving any other standard or investigational agents are ineligible.
2. Patients with history or current evidence of the following conditions are excluded: neuromuscular disorder with associated elevated CK (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy), pancreatitis, retinal vein occlusion, uncontrolled HIV, or Hepatitis B/C. An exception will be made for (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months and for subjects with cleared HBV and HCV infections, who may enroll in the study.
3. Known hypersensitivity or contraindication to any component of binimetinib or encorafenib or their excipients
4. Current use of a prohibited medication (including herbal medications, supplements, or foods), or use of a prohibited medication ≤ 7 days prior to the start of study treatment.
5. Patient has not recovered to ≤ Grade 1 non-hematologic toxic effects of prior therapy before starting study treatment. Note: Stable chronic conditions (≤ Grade 2) that are not expected to resolve (such as neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies) are exceptions and may enroll.
6. Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

   * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) ≤ 180 days prior to start date;
   * Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2);
   * Left ventricular ejection fraction (LVEF) < 50% as determined by MUGA or ECHO;
   * Uncontrolled hypertension defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy;
   * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
   * Triplicate average baseline QTc interval ≥ 480 ms.
7. Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (≤ 90 days) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs.
8. History of recent (≤ 90 days) thromboembolic or cerebrovascular event such as transient ischemic attack, cerebrovascular accident, or hemodynamically significant (massive or sub-massive) deep vein thrombosis or pulmonary emboli (DVT/PE). Note: Patients with DVT/PE that does not result in hemodynamic instability may enroll as long as they are anticoagulated for at least 4 weeks. Note: Patients with DVT/PE related to indwelling catheters or other procedures may enroll.
9. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible.
10. Pregnant women are excluded from this study because the effects of encorafenib and/or binimetinib on a fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with encorafenib or binimetinib, breastfeeding should be discontinued if the mother is treated with encorafenib and/or binimetinib.
11. Patients who previously received BRAF or MEK inhibitors are excluded (including but not limited to dabrafenib, vemurafenib, encorafenib, sorafenib, trametinib, binimetinib, cobimetinib, or selumetinib).
12. Patients will be excluded if their tumor harbors a known RAS activating mutation. This does not need to be specifically tested for eligibility.

3.4 Additional Inclusion Criteria for Surgical Arm

Patients must meet the above inclusion / exclusion criteria for consideration with one exception. Patients with a BRAF-V600 E or K mutated low-grade glioma for whom there is a strong clinical suspicion of progression to high-grade would also be eligible for this arm. Additionally:

1. Patients must have a clinical indication for a tumor surgery.
2. No a priori contraindication to biospecimen collection (blood, tumor, CSF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karisa C Schreck, MD, Principal Investigator — ABTC; Stuart A Grossman, MD, Study Chair — ABTC
Locations (3):
- United States (3):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued January 2020 -April 30 2022. The trial terminated early due to mandated closed to accrual for all ABTC studies as of 4/30/21. ABTC is closed to accrual and treatment on October 31 2023. The final trial clinical data includes a total of 5 subjects enrolled into the trial. Per original trial design, 56 subjects were required for the primary objective of the trial. The termination of the trial is considered an administrative termination.
Pre-assignment Details: 1 patient on Treatment Cohort 2 anaplastic PXAs was still on treatment at the time of the mandated stop of treating patients by NCI/CTEP. This patient continues to receive treatment but not on this study.
Groups:
- Treatment Cohort 1 AA & GBM; Treatment Cohort 2 Anaplastic PXAs; Treatment Cohort 3 Other Tumors: Encorafenib 450mg QD Binimetinib 45mg BID 28 day cycle
  Research Bloods
  Encorafenib: 450mg QD 28 day cycle
  Binimetinib: 45mg BID 28 day cycle
  Research Bloods: Baseline; pre-cycle 3; Pre-cycle 7; off Treatment
  Tumor Tissue: at time of surgery contrast enhancing and non enhancing tumor; 20 unstained slides
- Surgical Arm: Pre-op -14 days: Encorafenib 450mg QD and Binimetinib 45mg BID last dose of both drugs 2hrs prior to surgery
  Tumor; research blood; CSF samples
  post surgery: Encorafenib 450mg QD Binimetinib 45mg BID 28 day cycle
  Encorafenib: 450mg QD 28 day cycle
  Binimetinib: 45mg BID 28 day cycle
  Research Bloods: Baseline; pre-cycle 3; Pre-cycle 7; off Treatment
  Tumor Tissue: at time of surgery contrast enhancing and non enhancing tumor; 20 unstained slides
Period: Overall Study
Arm/Group | Treatment Cohort 1 AA & GBM | Treatment Cohort 2 Anaplastic PXAs | Surgical Arm | Treatment Cohort 3 Other Tumors
Started | 2 | 2 | 0 | 1
Completed | 2 | 1 | 0 | 0
Not Completed | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — pt had to stop treatment on this study but continued treatment off this study | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patient were enrolled on the Surgical arm. this study was terminated early by a mandate from NCI to shut down the ABTC Consortium due to wanting a different strategy for Brain Tumor Research. As such,
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Cohort 1 AA & GBM | Treatment Cohort 2 Anaplastic PXAs | Surgical Arm | Treatment Cohort 3 Other Tumors | Total
Number analyzed (Participants) | 2 | 2 | 0 | 1 | 5
Age, Continuous [Mean (Full Range); unit: years] | 30 [22 to 39] | 75 [27 to 77] |  | 26 [26 to 26] | 38 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 3
  Male | 1 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 2 | 1 | 0 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Karnofsky Performance Status Scale [Count of Participants; unit: Participants] — Higher score better "100 - Normal; no complaints; no evidence of disease; 90 - Able to carry on normal activity; minor signs or symptoms of disease, 80 - Normal activity with effort; some signs or symptoms of disease; 70 - Cares for self; unable to carry on normal activity or to do active work; 60 - Requires occasional assistance, but is able to care for most of his personal needs"
  Participants
    100-80 | 2 | 1 | 0 | 1 | 4
    70-60 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Radiographic Response Per RANO for 3 Treatment Cohorts
Description: Number of participants from each treatment cohort with response as defined by Response Assessment in Neuro-oncology (RANO) criteria: Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Stable Disease (SD)= <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Time Frame: Up to 1 year
Population: Due to early termination, results are given per cohort per patient, as the data is meaningless otherwise due to small numbers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cohort 1 AA & GBM | Treatment Cohort 2 Anaplastic PXAs | Treatment Cohort 3 Other Tumors
Number analyzed (Participants) | 2 | 2 | 1
Participants
  Complete Response (CR) | 0 | 1 | 0
  Partial Response (PR) | 2 | 0 | 0
  Stable Disease (SD) | 0 | 0 | 1
  Progression Disease (PD) | 0 | 1 | 0

2. Secondary Outcome: Progression Free Survival for 3 Treatment Cohorts
Description: Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status
Time Frame: up to 3 years
Population: Each row represents a specific patient. the number in that row equals the progression free survival for a specific patient, as there were only 5 patients
  Due to early termination, results are given per cohort per patient, as the data is meaningless otherwise due to small numbers
Measure: Number; unit: months
Arm/Group | Treatment Cohort 1 AA & GBM | Treatment Cohort 2 Anaplastic PXAs | Treatment Cohort 3 Other Tumors
Number analyzed (Participants) | 2 | 2 | 1
months
  pt 1: progression free survival: number analyzed (Participants) | 0 | 1 | 0
  pt 1: progression free survival |  | 33.5 |
  pt 2: progression free survival: number analyzed (Participants) | 0 | 1 | 0
  pt 2: progression free survival |  | 1.7 |
  pt 3: progression free survival: number analyzed (Participants) | 0 | 0 | 1
  pt 3: progression free survival |  |  | 4.2
  pt 4: progression free survival: number analyzed (Participants) | 1 | 0 | 0
  pt 4: progression free survival | 9.3 |  |
  pt 5: progression free survival: number analyzed (Participants) | 1 | 0 | 0
  pt 5: progression free survival | 10 |  |

3. Secondary Outcome: Overall Survival
Description: overall survival in months. Specific survival for each patient due to early termination
Time Frame: up to 3 years
Population: Due to early termination, results are given per cohort per patient, as the data is meaningless otherwise due to small numbers Each row represents a specific patient. the number in that row equals the overall survival for a specific patient, as there were only 5 patients
Measure: Number; unit: months
Arm/Group | Treatment Cohort 1 AA & GBM | Treatment Cohort 2 Anaplastic PXAs | Treatment Cohort 3 Other Tumors
Number analyzed (Participants) | 2 | 2 | 1
months
  pt number 1: number analyzed (Participants) | 0 | 1 | 0
  pt number 1 |  | 33.9 |
  pt number 2: number analyzed (Participants) | 0 | 1 | 0
  pt number 2 |  | 5.1 |
  pt number 3: number analyzed (Participants) | 0 | 0 | 1
  pt number 3 |  |  | 4.2
  pt number 4: number analyzed (Participants) | 1 | 0 | 0
  pt number 4 | 10.7 |  |
  pt number 5: number analyzed (Participants) | 1 | 0 | 0
  pt number 5 | 12.4 |  |

4. Secondary Outcome: Duration of Response - Complete and Partial
Description: Time from response to progression. Response is defined by RANO: Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Stable Disease (SD)= <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Time Frame: up to 3 year
Population: Each row represents the type of response. The number in that row equals the duration of response in months (mean) for all patients in cohort who had a response of the row title. There were 5 patients and only 3 patients had a response of CR or PR
Measure: Number; unit: months
Arm/Group | Treatment Cohort 1 AA & GBM | Treatment Cohort 2 Anaplastic PXAs | Treatment Cohort 3 Other Tumors
Number analyzed (Participants) | 2 | 2 | 1
months
  Duration of Complete response (CR) from base line in months: number analyzed (Participants) | 0 | 1 | 0
  Duration of Complete response (CR) from base line in months |  | 34 |
  Duration of Partial response (PR) from baseline months: number analyzed (Participants) | 1 | 1 | 0
  Duration of Partial response (PR) from baseline months | 8.5 | 8 |
  Duration of Progressive Disease (PD): number analyzed (Participants) | 1 | 0 | 1
  Duration of Progressive Disease (PD) | 2 |  | 4

5. Secondary Outcome: Number of Participants With Adverse Events as Defined by Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)
Description: time from first dose to 30 days post last dose
Time Frame: up to 3 years
Measure: Number; unit: percentage of patients
Groups:
- Patients Treated With Encorafenib or Binimetinib in All Cohorts: Toxicities with possible, or probable, or definite attribution to encorafenib or binimetinib, or both.
  Treatment Cohort 1 AA & GBM Treatment Cohort 2 anaplastic PXAs Treatment Cohort 3 Other Tumors
Arm/Group | Patients Treated With Encorafenib or Binimetinib in All Cohorts
Number analyzed (Participants) | 5
percentage of patients
  Dysphasia | 20
  alanine aminotransferase increased | 60
  anemia | 20
  blurred vision | 40
  CK serum | 20
  CPK increased | 60
  dysuria | 20
  fatigue | 20
  fever | 20
  floaters | 20
  insomnia | 20
  musculoskeletal, connective tissue disorder | 20
  myalgia | 20
  pain | 20
  right ciliorecinal artery occlusion | 20
  rash acneiform | 20
  retinopathy | 40
  urinary tract infection | 20
  vision decreased | 20
  weight gain | 20
  ASPARTATE AMINOTRANSFERASE INCREASED | 40

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Patients Treated With Encorafenib or Binimetinib in All Cohorts
All-Cause Mortality (participants affected / at risk) | 5/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Encorafenib or Binimetinib in All Cohorts (N=5)
CPK Increase (Investigations) | 1 (1)
eye disorder other (Eye disorders) | 1 (1) — RIGHT CILIORETINAL ARTERY OCCLUSION
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Encorafenib or Binimetinib in All Cohorts (N=5)
DYSPHASIA (Nervous system disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BLURRED VISION (Eye disorders) | 2 (2)
CK SERUM (Investigations) | 1 (1)
CPK INCREASED (Investigations) | 3 (3)
DYSURIA (Renal and urinary disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
FLOATERS (Eye disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
MUSCULOSKELETAL CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
RETINOPATHY (Eye disorders) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VISION DECREASED (Eye disorders) | 1 (1)
WEIGHT GAIN (Investigations) | 1 (1)
FEVER (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination, results are given per cohort per patient, as the data is meaningless otherwise due to small numbers.

The NCI/CTEP mandated the closure of ABTC Consortium and hence why this study was terminated early

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03973918/Prot_SAP_000.pdf